CLINICAL TRIAL: NCT01528345
Title: A Multicenter, Randomized, Double Blind, Placebo Controlled, Phase II Trial Evaluating the Safety and Efficacy of Dovitinib Combined With Fulvestrant, in Postmenopausal Patients With HER2- and HR+ Breast Cancer That Have Evidence of Disease Progression on or After Prior Endocrine Therapy
Brief Title: Trial Evaluating Dovitinib Combined With Fulvestrant, in Postmenopausal Patients With HER2- and HR+ Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow and low enrollment
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CTKI258A2210; 2011-001230-42 (EudraCT Number)
Record Dates: First submitted 2012-01-31; First posted 2012-02-08 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-05

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast Cancer; HER2-, HR+; post-menopausal; Locally advanced or metastatic Breast Cancer (HER2-, HR+)
MeSH Terms: conditions — Breast Neoplasms | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one; Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fulvestrant + Dovitinib active (Experimental): Fulvestrant in combination with the study drug Dovitinib.
  Interventions: Drug: Dovitinib; Drug: Fulvestrant
- Fulvestrant + Dovitinib placebo (Placebo Comparator): Fulvestrant in combination with a placebo matching Dovitinib.
  Interventions: Drug: Fulvestrant; Drug: Dovitinib Placebo

INTERVENTIONS:
Drug: Dovitinib — Active Dovitinib (in tablet form) taken orally at a dose of 500 mg (i.e., 5 x 100mg tablets) on a 5 days on/2 days off dosing schedule
  Other Names: TKI258
  Arms: Fulvestrant + Dovitinib active
Drug: Fulvestrant — Fulvestrant (in solution) injected intramuscularly at a dose of 500 mg once on Week 1 Day 1, Week 3 Day 1 and Week 5 Day 1 and subsequently once every 4 weeks on Day 1 of the week.
Drug: Dovitinib Placebo — Dovitinib Placebo (in tablet form) taken orally at a dose of 500 mg (i.e., 5 x 100mg tablets) on a 5 days on/2 days off dosing schedule
  Arms: Fulvestrant + Dovitinib placebo

SUMMARY:
This trial is designed to enroll postmenopausal patients with locally advanced or metastatic, HER2- and HR+ breast cancer not amenable to curative treatment by surgery or radiotherapy, and whose disease has progressed on or after prior endocrine therapy.

Patients must undergo molecular pre-screening prior to entry.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with HER2-, HR+ locally advanced or metastatic breast cancer
* Progression on or after endocrine treatment
* Measureable disease as per RECIST
* ECOG 0, 1 or 2

Exclusion Criteria:

* Evidence of CNS or leptomeningeal metastases
* Previous treatment with fulvestrant
* Previous chemotherapy for locally advanced or metastatic breast cancer
* Cirrhosis or chronic active/persistent hepatitis

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2012-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (63):
- United States (18):
  - Ironwood Cancer and Research Centers SC, Chandler, Arizona
  - Highlands Oncology Group Dept of Highlands Oncology Grp, Fayetteville, Arkansas
  - City of Hope National Medical Center COH 3, Duarte, California
  - University of California San Diego - Moores Cancer Center Moores UCSD Cancer Ctr. SC-1, La Jolla, California
  - Cedars Sinai Medical Center Samuel Oschin Cancer Center, Los Angeles, California
  - H. Lee Moffitt Cancer Center & Research Institute H. Lee Moffitt SC, Tampa, Florida
  - Oncology Specialists, SC Lutheran General Advanced Care, Park Ridge, Illinois
  - Indiana University Health Goshen Center for Cancer SC, Goshen, Indiana
  - Nebraska Methodist Hospital Estabrook Cancer Center, Omaha, Nebraska
  - Saint Barnabas Medical Center CancerCenter of Saint Barnabas, Livingston, New Jersey
  - ProHealth Care, Lake Success, New York
  - New York Oncology Hematology, P.C. Dept. of New York Oncology. PC, Troy, New York
  - Duke University Medical Center Duke (SC), Durham, North Carolina
  - Cancer Centers of the Carolinas Dept. of CC of the Carolinas, Greenville, South Carolina
  - Cancer Care Centers of South Texas / HOAST CCC of So. TX- San Antonio(2), San Antonio, Texas
  - Virginia Cancer Specialists, PC Dept.ofFairfax SC, Fairfax, Virginia
  - Medical Oncology Associates, PS, Spokane, Washington
  - Wenatchee Valley Medical Center Wenatchee Valley, Wenatchee, Washington
- Argentina (4):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Rio Negro, Viedma
- Austria (2):
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (2):
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Wilrijk
- Brazil (5):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Londrina, Paraná
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São José do Rio Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- France (6):
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Saint-Herblain Cédex
  - Novartis Investigative Site, Thonon-les-Bains
  - Novartis Investigative Site, Villejuif
- Hungary (5):
  - Novartis Investigative Site, Győr, Hungary
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Szolnok
- Italy (3):
  - Novartis Investigative Site, Macerata, MC
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Sondrio, SO
- Netherlands (2):
  - Novartis Investigative Site, Maastricht
  - Novartis Investigative Site, Rotterdam
- Novartis Investigative Site, Surquillo, Lima region, Peru
- Poland (3):
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Warsaw
- Russia (2):
  - Novartis Investigative Site, Ryazan, Russia
  - Novartis Investigative Site, Saint Petersburg
- South Africa (3):
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Parktown
  - Novartis Investigative Site, Port Elizabeth
- Spain (4):
  - Novartis Investigative Site, Toledo, Castille-La Mancha
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Valencia, Valencia
- Taiwan (3):
  - Novartis Investigative Site, Taichung, Taichung
  - Novartis Investigative Site, Niaosong Township, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan

REFERENCES:
- [Derived] Musolino A, Campone M, Neven P, Denduluri N, Barrios CH, Cortes J, Blackwell K, Soliman H, Kahan Z, Bonnefoi H, Squires M, Zhang Y, Deudon S, Shi MM, Andre F. Phase II, randomized, placebo-controlled study of dovitinib in combination with fulvestrant in postmenopausal patients with HR+, HER2- breast cancer that had progressed during or after prior endocrine therapy. Breast Cancer Res. 2017 Feb 10;19(1):18. doi: 10.1186/s13058-017-0807-8. PMID 28183331

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fulvestrant + Dovitinib Active | Fulvestrant + Dovitinib Placebo
Started | 47 | 50
Completed | 0 | 0
Not Completed | 47 | 50
Not completed — Adverse Event | 10 | 1
Not completed — Death | 1 | 1
Not completed — Non-compliance with study treatment | 1 | 0
Not completed — Progressive Disease | 26 | 40
Not completed — Study Terminated by Sponsor | 4 | 8
Not completed — Subject/Guardian Decision | 5 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): Consisted of all randomized patients. Following the intent-to-treat principle, patients were analyzed according to the treatment and stratum to which they were assigned at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fulvestrant + Dovitinib Active | Fulvestrant + Dovitinib Placebo | Total
Number analyzed (Participants) | 47 | 50 | 97
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.5 (9.02) | 61.7 (9.51) | 62.6 (9.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 50 | 97
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Based on Local Investigator Assessment
Description: PFS was defined as the time from the date of randomization to the date of the first radiologically documented disease progression or death due to any cause and was assessed based on RECIST v1.1. Responses include: Complete Response: Disappearance of all non-nodal target lesions; Partial Response: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters; Progressive Disease: At least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline; Stable Disease: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD; Unknown (UNK) Progression has not been documented and one or more target lesions have not been assessed or have been assessed using a different method than baseline.
Time Frame: Every 8 weeks assessed up to 34 months
Population: Full Analysis Set (FAS): Consisted of all randomized patients. Following the intent-to-treat principle, patients were analyzed according to the treatment and stratum to which they wereassigned at randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Fulvestrant + Dovitinib Active | Fulvestrant + Dovitinib Placebo
Number analyzed (Participants) | 47 | 50
Months
  All patients (n: 30, 34) | 5.5 [3.8 to 14.0] | 5.5 [3.5 to 10.7]
  FGF amplified patients (n: 9, 9) | 10.9 [3.5 to 16.5] | 5.5 [3.5 to 16.4]
  FGF non-amplified patients (n: 21, 25) | 5.5 [3.8 to 16.8] | 5.5 [1.9 to 12.8]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of patients with a best overall response of Complete Response (CR) or Partial Response (PR) as per RECIST v1.1. Responses include: Complete Response: Disappearance of all non-nodal target lesions; Partial Response: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters; Progressive Disease: At least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline; Stable Disease: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD; Unknown (UNK) Progression has not been documented and one or more target lesions have not been assessed or have been assessed using a different method than baseline.
Time Frame: Every 8 weeks assessed up to 34 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Fulvestrant + Dovitinib Active | Fulvestrant + Dovitinib Placebo
Number analyzed (Participants) | 47 | 50
Percentage of participants
  All patients | 27.7 [15.6 to 42.6] | 10.0 [3.3 to 21.8]
  FGF amplified patients | 20.0 [4.3 to 48.1] | 12.5 [1.6 to 38.3]
  FGF non-amplified patients | 31.3 [16.1 to 50.0] | 8.8 [1.9 to 23.7]

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as time from the date of the first documented response (CR or PR) to the date of the first documented or death due to disease. If a patient does not have a progression event, DOR will be censored on the date of the last adequate tumor assessment.
Time Frame: From date of first documented efficacy response (CR or PR) to time of documented progression (PD) whichever comes first, assessed up to 24 months
Population: This outcome measure was not analyzed as the study was terminated before duration of response could be analyzed.
Arm/Group | Fulvestrant + Dovitinib Active | Fulvestrant + Dovitinib Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Overall Survival (OS) Using Kaplan- Meier Method
Description: OS was defined as the time from the date of randomization to the date of death from any cause. If a patient is not known to have died at the date of analysis cut-off, the OS will be censored at the last date of contact.
Time Frame: From date of randomization to date of death from any cause whichever comes first, assessed up to 34 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Fulvestrant + Dovitinib Active | Fulvestrant + Dovitinib Placebo
Number analyzed (Participants) | 47 | 50
Months | NA [18.6 to NA] — N/A = Not estimable as there were too few events (not enough patients died by the data cutoff date for database lock). | 25.9 [18.4 to NA] — N/A = Not estimable as there were too few events (not enough patients died by the data cutoff date for database lock).

5. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety
Description: The type, frequency and severity of adverse events, laboratory values, and Electrocardiograms (ECGs) experienced by patients will be assessed according to Common Terminology Criteria for Adverse Events.
  The study enrollment was terminated early due to challenges in enrolling patients with FGF amplified status. See safety section for safety details.
Time Frame: Screening, Week 2, Week 4 and approximately every 4 weeks during treatment period (approximately 34 months)
Population: Safety Set: Consisted of all patients who received at least one dose of any compound of the study treatment (dovitinib +fulvestrant or placebo+fulvestrant). Patients were analyzed according to the actual study treatment received. Actual treatment received was defined as the treatment the patient received at the first day of study medication.
Measure: Number; unit: Participants
Arm/Group | Fulvestrant + Dovitinib Active | Fulvestrant + Dovitinib Placebo
Number analyzed (Participants) | 47 | 50
Participants | 47 | 50

6. Secondary Outcome: Time to Worsening of ECOG Performance Status
Description: Eastern Cooperative Oncology Group (ECOG) Performance Status (scales and criteria used by doctors and researchers to assess how a patient's disease is progressing and assess how the disease affects the daily living abilities of the patient.)
Time Frame: Screening, Every 4 weeks during treatment period, and every 8 weeks during follow-up (approximately 9-12 months)
Population: This outcome measure was not analyzed as the study was terminated before time to worsening ECOG performance could be analyzed.
Arm/Group | Fulvestrant + Dovitinib Active | Fulvestrant + Dovitinib Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Fulvestrant + Dovitinib Active | Fulvestrant + Dovitinib Placebo
Serious Adverse Events (participants affected / at risk) | 14/47 | 10/50
Other Adverse Events (participants affected / at risk) | 47/47 | 45/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant + Dovitinib Active (N=47) | Fulvestrant + Dovitinib Placebo (N=50)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 1
LUMBAR HERNIA (Gastrointestinal disorders) | 1 | 0
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
PANCREATITIS (Gastrointestinal disorders) | 0 | 1
VARICES OESOPHAGEAL (Gastrointestinal disorders) | 1 | 0
DEVICE BREAKAGE (General disorders) | 0 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 0
HYPERPYREXIA (General disorders) | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 1
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 0 | 1
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 | 0
INFECTION (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 0
TOOTH ABSCESS (Infections and infestations) | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
ISCHAEMIC CEREBRAL INFARCTION (Nervous system disorders) | 1 | 0
LARYNGOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 | 1
PIGMENTATION DISORDER (Skin and subcutaneous tissue disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 1
HYPOTENSION (Vascular disorders) | 0 | 1
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant + Dovitinib Active (N=47) | Fulvestrant + Dovitinib Placebo (N=50)
ANAEMIA (Blood and lymphatic system disorders) | 9 | 4
LEUKOPENIA (Blood and lymphatic system disorders) | 3 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 7 | 0
EAR PAIN (Ear and labyrinth disorders) | 5 | 0
VERTIGO (Ear and labyrinth disorders) | 6 | 0
DRY EYE (Eye disorders) | 5 | 0
LACRIMATION INCREASED (Eye disorders) | 6 | 0
VISION BLURRED (Eye disorders) | 3 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 4 | 3
ABDOMINAL PAIN (Gastrointestinal disorders) | 8 | 5
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 10 | 3
CONSTIPATION (Gastrointestinal disorders) | 8 | 5
DIARRHOEA (Gastrointestinal disorders) | 37 | 15
DRY MOUTH (Gastrointestinal disorders) | 5 | 1
DYSPEPSIA (Gastrointestinal disorders) | 12 | 0
GASTRITIS (Gastrointestinal disorders) | 3 | 0
NAUSEA (Gastrointestinal disorders) | 34 | 11
STOMATITIS (Gastrointestinal disorders) | 10 | 2
VOMITING (Gastrointestinal disorders) | 27 | 4
ASTHENIA (General disorders) | 18 | 11
FATIGUE (General disorders) | 16 | 13
INFLUENZA LIKE ILLNESS (General disorders) | 3 | 2
MALAISE (General disorders) | 4 | 1
OEDEMA PERIPHERAL (General disorders) | 3 | 3
PAIN (General disorders) | 4 | 0
PYREXIA (General disorders) | 6 | 5
CONJUNCTIVITIS (Infections and infestations) | 3 | 3
NASOPHARYNGITIS (Infections and infestations) | 3 | 1
URINARY TRACT INFECTION (Infections and infestations) | 2 | 4
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 15 | 5
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 10 | 4
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 11 | 1
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 9 | 4
LIPASE INCREASED (Investigations) | 3 | 3
WEIGHT DECREASED (Investigations) | 7 | 3
WEIGHT INCREASED (Investigations) | 1 | 3
DECREASED APPETITE (Metabolism and nutrition disorders) | 13 | 8
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 3 | 2
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 8 | 1
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 3 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7 | 9
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 | 9
BONE PAIN (Musculoskeletal and connective tissue disorders) | 3 | 4
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 3 | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 4 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 4 | 3
MYALGIA (Musculoskeletal and connective tissue disorders) | 5 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 9 | 3
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 3 | 1
AGEUSIA (Nervous system disorders) | 3 | 0
DIZZINESS (Nervous system disorders) | 4 | 2
DYSGEUSIA (Nervous system disorders) | 15 | 1
HEADACHE (Nervous system disorders) | 17 | 3
PARAESTHESIA (Nervous system disorders) | 2 | 3
SYNCOPE (Nervous system disorders) | 5 | 0
INSOMNIA (Psychiatric disorders) | 6 | 4
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 | 6
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 8 | 6
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 4 | 1
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 3 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 9 | 2
PRURITUS (Skin and subcutaneous tissue disorders) | 3 | 2
RASH (Skin and subcutaneous tissue disorders) | 16 | 3
HOT FLUSH (Vascular disorders) | 4 | 3
HYPERTENSION (Vascular disorders) | 13 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.